CLINICAL TRIAL: NCT01801111
Title: An Open-Label, Non-Randomized, Multicenter Phase I/II Trial of RO5424802 Given Orally to Non-Small Cell Lung Cancer Patients Who Have ALK Mutation and Who Have Failed Crizotinib Treatment
Brief Title: A Study of Alectinib (RO5424802) in Participants With Non-Small Cell Lung Cancer Who Have Anaplastic Lymphoma Kinase (ALK) Mutation and Failed Crizotinib Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP28673; 2012-004455-36 (EudraCT Number)
Record Dates: First submitted 2013-02-20; First posted 2013-02-28 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; alectinib

ARMS (1):
- Alectinib (Experimental): Participants will receive alectinib treatment continuously starting from Day 1 Cycle 1 (in 28-day cycles) until disease progression, death, or withdrawal for any other reasons, whichever occurs first. After PD, participants without EGFR mutation will continue treatment with alectinib alone and participants with EGFR mutation will receive alectinib in combination with erlotinib as per discretion of the treating physician.
  Interventions: Drug: Erlotinib; Drug: Alectinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib will be administered at a dose of 100 mg via tablet, orally, once daily in combination with alectinib to participants who progressed on alectinib alone treatment as per treating physician discretion.
  Other Names: Tarceva
Drug: Alectinib — Alectinib will be administered at a dose of 600 milligrams (mg) via capsule, orally, twice daily.
  Other Names: RO5452802

SUMMARY:
This open-label, non-randomized, multicenter, Phase 1/2 study will evaluate the safety and efficacy of alectinib in participants with non-small cell lung cancer who have ALK mutation and failed crizotinib treatment. In Part 1, cohorts of participants will receive escalating doses of alectinib orally twice daily. In Part 2, participants will receive the recommended phase 2 dose (RP2D) of alectinib as determined in Part 1. Treatment will continue in Part 1 and Part 2 on the same dose until disease progression. In Part 3, following disease progression, participants without epidermal growth factor receptor (EGFR) mutation will be offered continued treatment with alectinib, participants with EGFR mutations will be offered a combination of alectinib and erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic non-small cell lung cancer (stage IIIB or IV by American Joint Committee on Cancer [AJCC])
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Documented ALK rearrangement based on Food and Drug Administration (FDA)-approved test
* Prior treatment with crizotinib and progression according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1) criteria. Participants had to have a minimum 1-week wash-out period between the last dose of crizotinib and the first dose of study treatment. Participants can either be chemotherapy-naïve or have received at least one line of platinum-based chemotherapy
* Adequate hematologic, hepatic, and renal function
* Participants with brain or leptomeningeal metastases are allowed if protocol defined criteria are met
* Measurable disease according to RECIST v1.1 prior to administration of first dose of study drug

Exclusion Criteria:

* Receipt of any other ALK inhibitors in addition to crizotinib
* Receipt of any prior cytotoxic chemotherapy for ALK-positive NSCLC within 4 weeks prior to the first dose of study drug
* Participants who received crizotinib or any other tyrosine kinase inhibitors need to have a minimum 1-week washout period before the first dose of study drug
* Active or uncontrolled infectious diseases requiring treatment
* National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (NCI CTCAE v4.03) Grade 3 or higher toxicities due to prior therapy that have not shown improvement and are considered to interfere with current study medication
* History of organ transplant
* Co-administration of anti-cancer therapies other than those administered in this study
* Baseline corrected Q-T interval (QTc) greater than (>) 470 milliseconds, or baseline symptomatic bradycardia (less than 45 heart beats per minute)
* Pregnant or breastfeeding women
* Known Human Immunodeficiency Virus (HIV) positivity or Acquired Immunodeficiency Syndrome (AIDS)-related illness
* History of hypersensitivity to any of the additives in the alectinib formulation
* Any clinically significant concomitant disease or condition that could interfere with, or for which treatment might interfere with, the conduct of the study, or absorption of oral medications, or that would, in the opinion of the principal investigator, pose an unacceptable risk to the participant in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2014-10-24 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (84):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Jude Heritage Healthcare, Fullerton, California
  - UC Irvine Medical Center, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - UCLA Cancer Center; Premiere Oncology, A Medical Corporation, Santa Monica, California
  - Advanced Medical Specialties, Miami, Florida
  - Florida Hospital Cancer Inst, Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Midwestern Regional Medical Center; Office of Research, Zion, Illinois
  - Washington University; Wash Uni. Sch. Of Med, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Columbia University Medical Center; Department of Hematology/Oncology, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Texas Oncology, P.A., Dallas, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Australia (3):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Townsville General Hospital, Douglas, Queensland
- Belgium (3):
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - AZ Delta (Campus Wilgenstraat), Roeselare
- University Hospital Herlev, Herlev, Denmark
- France (13):
  - CHU Angers - Hôpital Hôtel Dieu, Angers
  - Hopital Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Georges François Leclerc; Service Pharmacie, Bp 77980, Dijon
  - CHU de Grenoble - Hôpital Nord; Service d'Oncologie Thoracique, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hôpital Nord - AP-HM Marseille#; Gastroenterology and Hepatology, Marseille
  - Groupe Hospitalier Sud - Hôpital Haut Lévêque, Pessac
  - Hopital Pontchaillou - CHU de Rennes, Rennes
  - ICO Rene Gauducheau; CEC, Saint-Herblain
  - Nouvel Hopital Civil - CHU Strasbourg, Strasbourg
  - CHU de Toulouse - Hôpital Larrey, Toulouse
- Germany (6):
  - Charité Campus Virchow-Klinikum; Department of Cardiology, Berlin
  - Klinikum Koeln-Merheim, Cologne
  - Diakonie Kaiserswerth; Florence-Nightingale-Krankenhaus, Düsseldorf
  - LungenClinic Großhansdorf, Großhansdorf
  - Lungenklinik Hemer, Hemer
  - Mathias-Spital Rheine, Rheine
- Italy (11):
  - A.O. Universitaria Di Parma, Parma, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO), Aviano, Friuli Venezia Giulia
  - Istituto Nazionale Tumori Regina Elena IRCCS, Rome, Lazio
  - AO San Camillo Forlanini, Rome, Lazio
  - Ospedale San Raffaele, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Niguarda (Ospedale Niguarda Ca' Granda), Milan, Lombardy
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Ospedale Versilia, Lido di Camaiore, Tuscany
  - Presidio Ospedaliero Campo di Marte, Lucca, Tuscany
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia, Umbria
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Netherlands (3):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Maastricht University Medical Centre; Afdeling Klinische Farmacie en Toxicologie, Maastricht
- FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin"; Chemotherapy Departement, Moskva, Moscow Oblast, Russia
- Singapore (2):
  - National University Hospital; Investigational Medicine Unit, Singapore
  - Johns Hopkins Singapore, Singapore
- South Korea (6):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System; Pharmacy, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (10):
  - Hospital General Univ. de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitario Quiron Dexeus, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hosp Clinico Univ Lozano Blesa, Zaragoza
- Karolinska, Stockholm, Sweden
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung Univ Hosp, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal Marsden Hospital;Dept of Haematology Oncology Research, London
  - Royal Marsden Hospital - London, London

REFERENCES:
- [Derived] Ou SI, Gadgeel SM, Barlesi F, Yang JC, De Petris L, Kim DW, Govindan R, Dingemans AM, Crino L, Lena H, Popat S, Ahn JS, Dansin E, Mitry E, Muller B, Bordogna W, Balas B, Morcos PN, Shaw AT. Pooled overall survival and safety data from the pivotal phase II studies (NP28673 and NP28761) of alectinib in ALK-positive non-small-cell lung cancer. Lung Cancer. 2020 Jan;139:22-27. doi: 10.1016/j.lungcan.2019.10.015. Epub 2019 Oct 14. PMID 31706099
- [Derived] Morcos PN, Nueesch E, Jaminion F, Guerini E, Hsu JC, Bordogna W, Balas B, Mercier F. Exposure-response analysis of alectinib in crizotinib-resistant ALK-positive non-small cell lung cancer. Cancer Chemother Pharmacol. 2018 Jul;82(1):129-138. doi: 10.1007/s00280-018-3597-5. Epub 2018 May 10. PMID 29748847
- [Derived] Gadgeel SM, Shaw AT, Govindan R, Gandhi L, Socinski MA, Camidge DR, De Petris L, Kim DW, Chiappori A, Moro-Sibilot DL, Duruisseaux M, Crino L, De Pas T, Dansin E, Tessmer A, Yang JC, Han JY, Bordogna W, Golding S, Zeaiter A, Ou SI. Pooled Analysis of CNS Response to Alectinib in Two Studies of Pretreated Patients With ALK-Positive Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Dec;34(34):4079-4085. doi: 10.1200/JCO.2016.68.4639. Epub 2016 Oct 31. PMID 27863201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall study status was confirmed as completed. Here, 'study terminated by sponsor' in reason for study not completed means participants were transitioned to commercial supply of alectinib (where it was available) or transitioned to a roll-over study BO39694 (NCT03194893) where they continued to receive alectinib treatment.
Pre-assignment Details: Part 1 of study was planned to determine recommended Phase 2 dose (RP2D) of alectinib to be used in Part 2. During the conduct of Part 1 for this study, RP2D was confirmed in Study NP28761 (NCT01871805). Hence Part 1 participants were merged into Part 2. Part 3 was post-progression treatment period.
Groups:
- Alectinib: Participants received alectinib at a dose of 600 milligrams (mg) via capsule, orally, twice daily, continuously starting on Day 1 Cycle 1 (in 28-day cycles) until disease progression (PD), death, or withdrawal for any other reasons, whichever occurred first. After PD, participants were allowed to continue treatment with alectinib as per the discretion of the treating physician.
Period: Overall Study
Arm/Group | Alectinib
Started | 138
Completed | 0
Not Completed | 138
Not completed — Adverse Event | 12
Not completed — Death | 8
Not completed — Physician Decision | 5
Not completed — Other | 1
Not completed — Withdrawal by Subject | 4
Not completed — Study Terminated by Sponsor | 27
Not completed — Progressive Disease | 81

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population, which included all participants who received at least one dose of alectinib.
Groups:
- Alectinib: Participants received alectinib at a dose of 600 mg via capsule, orally, twice daily, continuously starting on Day 1 Cycle 1 (in 28-day cycles) until PD, death, or withdrawal for any other reasons, whichever occurred first. After PD, participants were allowed to continue treatment with alectinib as per the discretion of the treating physician.
Arm/Group | Alectinib
Number analyzed (Participants) | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 61

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Alectinib
Description: RP2D was to be determined based on the safety and tolerability profile of the study treatment.
Time Frame: Cycle 1 (up to 28 days)
Population: The endpoint was not analyzed in this study as the RP2D was confirmed in study NP28761 (NCT01871805).
Arm/Group | Alectinib
Number analyzed (Participants) | 0

2. Primary Outcome: Percentage of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were to be assessed based on the National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.3 (NCI-CTCAE v 4.3). DLTs: drug-related toxicities that meet any one of the following criteria: Grade 4 thrombocytopenia; Grade 3 thrombocytopenia with bleeding; Grade 4 neutropenia continuing for greater than or equal to (>/=) 7 consecutive days or neutropenic fever; Non-hematological toxicity of Grade 3 or higher; Adverse events that require interruption of treatment for a total of >/=7 days.
Time Frame: Cycle 1 (up to 28 days)
Population: The endpoint was not analyzed in this study as the RP2D was confirmed in study NP28761 (NCT01871805).
Arm/Group | Alectinib
Number analyzed (Participants) | 0

3. Primary Outcome: Percentage of Participants Achieving Objective Response (Complete Response [CR] or Partial Response [PR]) as Assessed by Independent Radiological Review Committee (IRC) in Response Evaluable (RE) Population
Description: Tumor response was assessed by IRC according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Objective response was defined as percentage of participants with a CR or PR that was confirmed by repeat assessments >/=4 weeks after initial documentation. CR was defined as disappearance of all target, non-target lesions; normalization of tumor marker level; and reduction in all lymph nodes size to less than (<) 10 millimeters (mm). PR was defined as >/=30 percent (%) decrease in the sum of diameters (SoD) of target lesions (taking as reference the baseline SoD). The 95% confidence interval (CI) was computed using Clopper-Pearson method.
Time Frame: Baseline; assessments every 8 weeks post-baseline until progressive disease, unacceptable toxicity, consent withdrawal, death, other reason deemed by investigator, or last tumor assessment (up to approximately 2.5 years)
Population: Analysis was performed on RE population (IRC) which included all participants with measurable disease at baseline according to the IRC, who had baseline tumor assessment and received at least one dose of alectinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 122
percentage of participants | 50.8 [41.62 to 59.98]
Statistical Analysis 1: Comparison: Alectinib; Tests null hypothesis that the objective response rate (ORR) is equal to 35% versus the alternative hypothesis that the objective response rate was not equal to 35%; Test type: Other; p = 0.0005, Exact Clopper-Pearson CI

4. Primary Outcome: Percentage of Participants Achieving Objective Response (CR or PR) as Assessed by IRC in Chemotherapy-Pretreated Participants
Description: Tumor response was assessed by IRC according to RECIST v1.1. Objective response was defined as percentage of participants with a CR or PR that was confirmed by repeat assessments >/=4 weeks after initial documentation. CR was defined as disappearance of all target, non-target lesions; normalization of tumor marker level; and reduction in all lymph nodes size to <10 mm. PR was defined as >/=30% decrease in the SoD of target lesions (taking as reference the baseline SoD). The 95% CI was computed using Clopper-Pearson method.
Time Frame: as for outcome 3
Population: Analysis was performed on RE population (IRC) participants who received prior chemotherapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 96
percentage of participants | 44.8 [34.63 to 55.29]
Statistical Analysis 1: Comparison: Alectinib; Tests null hypothesis that the ORR is equal to 35% versus the alternative hypothesis that the objective response rate was not equal to 35%; Test type: Other; p = 0.0599, Exact Clopper-Pearson CI

5. Secondary Outcome: Percentage of Participants Achieving Objective Response (CR or PR) as Assessed by IRC in Chemotherapy-Naive Participants
Description: Tumor response was assessed by IRC according to RECIST v1.1. Objective response was defined as percentage of participants with a CR or PR that was confirmed by repeat assessments >/=4 weeks after initial documentation. CR was defined as disappearance of all target, non-target lesions; normalization of tumor marker level; and reduction in all lymph nodes size to <10 mm. PR was defined as >/=30% decrease in the SoD of target lesions (taking as reference the baseline SoD).
Time Frame: as for outcome 3
Population: Analysis was performed on RE population (IRC) participants who did not receive prior chemotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 26
percentage of participants | 73.1

6. Secondary Outcome: Percentage of Participants Achieving Objective Response (CR or PR) as Assessed by Investigator in RE Population
Description: Tumor response was assessed by the investigator according to RECIST v1.1. Objective response was defined as percentage of participants with a CR or PR that was confirmed by repeat assessments >/=4 weeks after initial documentation. CR was defined as disappearance of all target, non-target lesions; normalization of tumor marker level; and reduction in all lymph nodes size to <10 mm. PR was defined as >/=30% decrease in the SoD of target lesions (taking as reference the baseline SoD). The 95% CI was computed using Clopper-Pearson method.
Time Frame: as for outcome 3
Population: Analysis was performed on RE population (Investigator) which included all participants with measurable disease at baseline according to the investigator, who had baseline tumor assessment and received at least one dose of alectinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 138
percentage of participants | 51.4 [42.80 to 60.04]
Statistical Analysis 1: Comparison: Alectinib; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.0001, Exact Clopper-Pearson CI

7. Secondary Outcome: Percentage of Participants Achieving Objective Response (CR or PR) as Assessed by Investigator in Chemotherapy-Pretreated Participants
Description: Tumor response was assessed by the investigator according to RECIST v1.1. Objective response was defined as percentage of participants with a CR or PR that was confirmed by repeat assessments >/=4 weeks after initial documentation. CR was defined as disappearance of all target, non-target lesions; normalization of tumor marker level; and reduction in all lymph nodes size to <10 mm. PR was defined as >/=30% decrease in the SoD of target lesions (taking as reference the baseline SoD).
Time Frame: as for outcome 3
Population: Analysis was performed on RE population (investigator) participants who received prior chemotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 110
percentage of participants | 50.0

8. Secondary Outcome: Percentage of Participants Achieving Objective Response (CR or PR) as Assessed by Investigator in Chemotherapy-Naive Participants
Description: as for outcome 7
Time Frame: as for outcome 3
Population: Analysis was performed on RE population (investigator) participants who did not receive prior chemotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 28
percentage of participants | 57.1

9. Secondary Outcome: Duration of Response (DoR) as Assessed by IRC in RE Population
Description: DoR was defined as the time from the first observation of an objective tumor response (CR or PR) until first observation of progressive disease (PD) according to RECIST v1.1 or death from any cause. CR: disappearance of all target, non-target lesions; normalization of tumor marker level; and reduction in all lymph nodes size to <10 mm. PR: >/=30% decrease in the SoD of target lesions (taking as reference the baseline SoD). PD: >/=20% relative increase and >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-target lesions. Duration of response was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley. Participants who did not progress or die after a confirmed objective response were censored at the date of their last tumor assessment.
Time Frame: as for outcome 3
Population: Analysis was performed on RE population (IRC) participants with documented objective response as assessed by IRC according to RECIST v1.1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib
Number analyzed (Participants) | 62
months | 15.2 [11.2 to 24.9]

10. Secondary Outcome: Percentage of Participants With PD as Assessed by IRC According to RECIST v1.1 or Death From Any Cause in Safety Population
Description: According to RECIST v1.1, PD was defined as >/=20% relative increase and >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-target lesions.
Time Frame: as for outcome 3
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 138
percentage of participants | 71.0

11. Secondary Outcome: Progression Free Survival (PFS) as Assessed by IRC in Safety Population
Description: PFS was defined as the time interval between the date of the first treatment and the date of PD or death from any cause, whichever occurred first. PD: >/=20% relative increase and >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-target lesions. PFS was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley. Participants who neither progressed nor died at the time of assessment or who were lost to follow-up were censored at the date of the last tumor assessment. Participants with no post-baseline assessments were censored at the date of first dose.
Time Frame: as for outcome 3
Population: Analysis was performed on safety population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib
Number analyzed (Participants) | 138
months | 8.9 [5.6 to 12.8]

12. Secondary Outcome: Percentage of Participants Who Died of Any Cause
Description: Percentage of participants who died of any cause was reported.
Time Frame: Baseline up to death from any cause (up to approximately 4 years)
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 138
percentage of participants | 54.3

13. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first treatment to the date of death, regardless of the cause of death. OS was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley. Participants who did not die were censored at the date last known to be alive.
Time Frame: Baseline up to death from any cause (up to approximately 4 years)
Population: Analysis was performed on safety population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib
Number analyzed (Participants) | 138
months | 29.2 [21.5 to 44.4]

14. Secondary Outcome: Percentage of Participants Achieving CR, PR or Stable Disease (SD) According to RECIST v1.1 in RE Population
Description: The disease control rate (DCR) was defined as the percentage of participants achieving CR, PR, or SD that lasted for at least 16 weeks. Tumor response was assessed by the investigator and IRC according to RECIST v1.1. CR: disappearance of all target, non-target lesions; normalization of tumor marker level; and reduction in all lymph nodes size to <10 mm. PR: >/=30% decrease in the SoD of target lesions (taking as reference the baseline SoD). PD: >/=20% relative increase and >/=5 mm of absolute increase in the SoD, taking as reference the smallest SoD recorded since treatment started; 1 or more new lesion(s); and/or unequivocal progression of non-target lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SoD while on study. The 95% CI was computed using Clopper-Pearson method.
Time Frame: as for outcome 3
Population: Analysis was performed on RE population which included all participants with measurable disease at baseline, who had baseline tumor assessment, and who received at least one dose of alectinib. Here, 'Number Analyzed'=number of participant evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 138
percentage of participants
  IRC Assessment: number analyzed (Participants) | 122
  IRC Assessment | 63.9 [54.75 to 72.43]
  Investigator Assessment | 69.6 [61.16 to 77.11]

15. Secondary Outcome: Percentage of Participants Achieving Central Nervous System (CNS) Objective Response as Assessed by IRC According to RECIST v1.1
Description: CNS response was assessed by IRC according to RECIST v1.1. CNS Objective response was defined as percentage of participants with a CR or PR. CR was defined as disappearance of all CNS lesions. PR was defined as >/=30% decrease in the SoD of measurable CNS lesions (taking as reference the baseline SoD). The 95% CI was computed using Clopper-Pearson method.
Time Frame: as for outcome 3
Population: Analysis was performed on safety population participants with measurable CNS lesions at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 34
percentage of participants | 58.8 [40.70 to 75.35]

16. Secondary Outcome: Percentage of Participants Achieving CNS Objective Response as Assessed by IRC According to Radiology Assessment in Neuro-Oncology (RANO) Criteria
Description: CNS response was assessed by IRC according to RANO criteria. CNS Objective response: percentage of participants with a CR or PR that was confirmed by repeat assessments >/=4 weeks after initial documentation. CR was defined as complete disappearance of all enhancing measurable, non-measurable disease; stable or improved non-enhancing lesions; no new lesions; no corticosteroids (or only physiologic replacement dose), and clinically stable or improved. PR was defined as >/=50% decrease compared to screening in the sum of the products of the diameters (SPD) of enhancing measurable lesions; no progression of non-measurable disease (enhancing and non-enhancing lesions); no new lesions; no corticosteroids (or only physiologic replacement dose), and clinically stable or improved. The 95% CI was computed using Clopper-Pearson method.
Time Frame: Baseline; assessments every 8 weeks post-baseline until progressive disease, unacceptable toxicity, consent withdrawal, death, other reason deemed by investigator; then survival follow-up until cutoff 18 August 2014 (up to approximately 53 weeks)
Population: Analysis was performed on safety population participants with measurable CNS lesions at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 34
percentage of participants | 44.1 [27.19 to 62.11]

17. Secondary Outcome: CNS Duration of Response (CDoR) as Assessed by IRC According to RECIST v1.1
Description: CDoR was defined as the time from the first observation of a CNS objective response (CR or PR) until first observation of CNS progression as assessed by IRC according to RECIST v 1.1 or death from any cause. CR: disappearance of all CNS lesions. PR: >/=30% decrease in the SoD of measurable CNS lesions (taking as reference the baseline SoD). CNS progression: >/=20% increase in the SoD of measurable CNS lesions (with an absolute increase of at least 5 mm), taking as reference the baseline SoD; 1 or more new CNS lesion(s); and/or unequivocal progression of non-measurable CNS lesions. CDoR was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 3
Population: Analysis was performed on safety population participants with measurable CNS lesions at baseline and who had CNS objective response as assessed by IRC according to RECIST v1.1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib
Number analyzed (Participants) | 20
months | 11.1 [7.1 to NA] — The upper limit of 95% CI could not be estimated due to high number of censored participants.

18. Secondary Outcome: CDoR as Assessed by IRC According to RANO Criteria
Description: CDoR: time from the CNS objective response until CNS progression as assessed by IRC according to RANO criteria or death from any cause. CR: complete disappearance of all enhancing measurable, non-measurable disease; stable/improved non-enhancing lesions; no new lesions; no corticosteroids, and clinically stable/improved. PR: >/=50% decrease compared to screening in SPD of enhancing measurable lesions; no progression of non-measurable disease; no new lesions; no corticosteroids, and clinically stable/improved. Progression: >/=25% increase in SPD of enhancing measurable lesions compared to best response on study; stable/increasing doses of corticosteroids; significant increase in non-enhancing lesions not caused by co-morbid events; any new lesions; progression of non-measurable disease; or clinical deterioration not attributable to other non-tumor causes. CDoR was estimated by Kaplan-Meier method and 95% CI was assessed using method of Brookmeyer and Crowley.
Time Frame: as for outcome 16
Population: Analysis was performed on safety population participants with measurable CNS lesions at baseline and who had CNS objective response as assessed by IRC according to RANO criteria.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib
Number analyzed (Participants) | 15
months | 7.6 [7.4 to 7.6]

19. Secondary Outcome: Percentage of Participants With CNS Progression as Assessed by IRC According to RECIST v 1.1
Description: According to RECIST v 1.1, CNS progression was defined as >/=20% increase in the SoD of measurable CNS lesions (with an absolute increase of at least 5 mm), taking as reference the baseline SoD; 1 or more new CNS lesion(s); and/or unequivocal progression of non-measurable CNS lesions.
Time Frame: as for outcome 16
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Alectinib
Number analyzed (Participants) | 138
percentage of participants | 18.8

20. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Alectinib
Description: Cmax for alectinib was estimated from plasma concentration versus time data by non-compartmental methods of analysis using Phoenix WinNonlin v6.2 (Pharsight Corporation) software.
Time Frame: Pre-dose (0 hours [hrs]), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: Analysis was performed on Pharmacokinetic (PK) Evaluable Population, which included all participants who received any dose of alectinib and who had at least one post-baseline PK sample available. Here, 'Number Analyzed'=number of participant evaluable for specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Alectinib
Number analyzed (Participants) | 28
nanograms per milliliter (ng/mL)
  Day 1 | 204 (47.6)
  Day 21: number analyzed (Participants) | 26
  Day 21 | 933 (34.8)

21. Secondary Outcome: Time to Cmax (Tmax) of Alectinib
Description: Tmax for alectinib was estimated from plasma concentration versus time data by non-compartmental methods of analysis using Phoenix WinNonlin v6.2 software.
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: Analysis was performed on PK Evaluable Population. Here, 'Number Analyzed'=number of participant evaluable for specified category.
Measure: Median (Full Range); unit: hrs
Arm/Group | Alectinib
Number analyzed (Participants) | 28
hrs
  Day 1 | 5.89 [2.00 to 10.00]
  Day 21: number analyzed (Participants) | 26
  Day 21 | 4.12 [0.0 to 11.18]

22. Secondary Outcome: Time to Last Measurable Plasma Concentration (Tlast) of Alectinib
Description: Tlast for alectinib was estimated from plasma concentration versus time data by non-compartmental methods of analysis using Phoenix WinNonlin v6.2 software.
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hrs
Arm/Group | Alectinib
Number analyzed (Participants) | 28
hrs
  Day 1 | 11.59 (3.9)
  Day 21: number analyzed (Participants) | 26
  Day 21 | 11.65 (3.8)

23. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 10 Hours Post-dose (AUC[0-10]) of Alectinib
Description: The AUC(0-10) of alectinib was calculated using the linear trapezoidal rule and actual sampling times (with the exception of pre-dose which was set to zero).
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hrs*nanograms per milliliter (hrs*ng/mL)
Arm/Group | Alectinib
Number analyzed (Participants) | 28
hrs*nanograms per milliliter (hrs*ng/mL)
  Day 1 | 1140 (44.5)
  Day 21: number analyzed (Participants) | 26
  Day 21 | 7860 (37.2)

24. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Tlast (AUC[0-last]) of Alectinib
Description: The AUC(0-last) of alectinib was calculated using the linear trapezoidal rule and actual sampling times (with the exception of pre-dose which was set to zero).
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hrs*ng/mL
Arm/Group | Alectinib
Number analyzed (Participants) | 28
hrs*ng/mL
  Day 1 | 1340 (44.9)
  Day 21: number analyzed (Participants) | 26
  Day 21 | 9090 (36.9)

25. Secondary Outcome: Cmax of Alectinib Metabolite
Description: Cmax for alectinib metabolite was estimated from plasma concentration versus time data by non-compartmental methods of analysis using Phoenix WinNonlin v6.2 software.
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Alectinib
Number analyzed (Participants) | 28
nanograms per milliliter (ng/mL)
  Day 1 | 57.2 (68.6)
  Day 21: number analyzed (Participants) | 26
  Day 21 | 303 (33.5)

26. Secondary Outcome: Tmax of Alectinib Metabolite
Description: Tmax for alectinib metabolite was estimated from plasma concentration versus time data by non-compartmental methods of analysis using Phoenix WinNonlin v6.2 software.
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 21
Measure: Median (Full Range); unit: hrs
Arm/Group | Alectinib
Number analyzed (Participants) | 28
hrs
  Day 1 | 8.03 [5.97 to 11.18]
  Day 21: number analyzed (Participants) | 26
  Day 21 | 7.00 [0.0 to 12.00]

27. Secondary Outcome: Tlast of Alectinib Metabolite
Description: Tlast for alectinib metabolite was estimated from plasma concentration versus time data by non-compartmental methods of analysis using Phoenix WinNonlin v6.2 software.
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hrs
Arm/Group | Alectinib
Number analyzed (Participants) | 28
hrs
  Day 1 | 11.59 (3.9)
  Day 21: number analyzed (Participants) | 26
  Day 21 | 11.65 (3.8)

28. Secondary Outcome: AUC(0-10) of Alectinib Metabolite
Description: The AUC(0-10) of alectinib metabolite was calculated using the linear trapezoidal rule and actual sampling times (with the exception of pre-dose which was set to zero).
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hrs*ng/mL
Arm/Group | Alectinib
Number analyzed (Participants) | 28
hrs*ng/mL
  Day 1 | 300 (68.4)
  Day 21: number analyzed (Participants) | 26
  Day 21 | 2590 (35.0)

29. Secondary Outcome: AUC(0-last) of Alectinib Metabolite
Description: The AUC(0-last) of alectinib metabolite was calculated using the linear trapezoidal rule and actual sampling times (with the exception of pre-dose which was set to zero).
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hrs*ng/mL
Arm/Group | Alectinib
Number analyzed (Participants) | 28
hrs*ng/mL
  Day 1 | 378 (67.5)
  Day 21: number analyzed (Participants) | 26
  Day 21 | 3040 (34.9)

30. Secondary Outcome: Metabolite to Parent Ratio Based on AUC(0-10)
Description: Metabolite to parent ratio based on AUC(0-10) was computed as AUC(0-10) of metabolite divided by AUC(0-10) of parent drug (alectinib) corrected for the molecular weight of parent divided by the molecular weight of the metabolite.
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Alectinib
Number analyzed (Participants) | 28
Ratio
  Day 1 | 0.278 (41.0)
  Day 21: number analyzed (Participants) | 26
  Day 21 | 0.349 (28.7)

31. Secondary Outcome: Metabolite to Parent Ratio Based on AUC(0-last)
Description: Metabolite to parent ratio based on AUC(0-last) was computed as AUC(0-last) of metabolite divided by AUC(0-last) of parent drug (alectinib) corrected for the molecular weight of parent divided by the molecular weight of the metabolite.
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hrs post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Alectinib
Number analyzed (Participants) | 28
Ratio
  Day 1 | 0.298 (41.2)
  Day 21: number analyzed (Participants) | 26
  Day 21 | 0.354 (28.7)

32. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Alectinib
Time Frame: Pre-dose (0 hrs) on Day 21 of Cycle 1
Population: Analysis was performed on PK Evaluable Population. Here, 'Overall Number of Participants Analyzed'=number of participant evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alectinib
Number analyzed (Participants) | 26
ng/mL | 761 (42.9)

33. Secondary Outcome: Ctrough of Alectinib Metabolite
Time Frame: Pre-dose (0 hrs) on Day 21 of Cycle 1
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alectinib
Number analyzed (Participants) | 26
ng/mL | 244 (37.8)

34. Secondary Outcome: Peak to Trough Ratio of Alectinib
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hours post-dose on Day 21 of Cycle 1
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Alectinib
Number analyzed (Participants) | 26
Ratio | 1.23 (14.4)

35. Secondary Outcome: Accumulation Ratio of Alectinib
Description: Accumulation ratio after repeat dosing was computed as AUC(0-10) on Day 21 divided by AUC(0-10) on Day 1.
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hours post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Alectinib
Number analyzed (Participants) | 26
Ratio | 6.95 (42.1)

36. Secondary Outcome: Accumulation Ratio of Alectinib Metabolite
Description: Accumulation ratio after repeat dosing was computed as AUC(0-10) on Day 21 divided by AUC(0-10) on Day 1.
Time Frame: Pre-dose (0 hrs), and 0.5, 1, 2, 4, 6, 8, 10, 12 hours post-dose on Day 1 and Day 21 of Cycle 1
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Alectinib
Number analyzed (Participants) | 26
Ratio | 8.68 (64.2)

ADVERSE EVENTS:
Time Frame: From Baseline until 28 days after the last dose of study drug (overall up to approximately 4 years)
Description: Analysis was performed on safety population.
Arm/Group | Alectinib
All-Cause Mortality (participants affected / at risk) | 75/138
Serious Adverse Events (participants affected / at risk) | 39/138
Other Adverse Events (participants affected / at risk) | 133/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alectinib (N=138)
Myocardial infarction (Cardiac disorders) | 1
Retinal detachment (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Appendicitis perforated (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Pleural infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Haemorrhage (Vascular disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
International normalised ratio increased (Investigations) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 2
Ureterolithiasis (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alectinib (N=138)
Anaemia (Blood and lymphatic system disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 17
Constipation (Gastrointestinal disorders) | 53
Diarrhoea (Gastrointestinal disorders) | 27
Nausea (Gastrointestinal disorders) | 32
Vomiting (Gastrointestinal disorders) | 22
Asthenia (General disorders) | 31
Fatigue (General disorders) | 43
Oedema (General disorders) | 9
Oedema peripheral (General disorders) | 42
Pyrexia (General disorders) | 17
Upper respiratory tract infection (Infections and infestations) | 21
Alanine aminotransferase increased (Investigations) | 15
Asparatate aminotransferase increased (Investigations) | 18
Blood bilirubin increased (Investigations) | 18
Decreased appetite (Metabolism and nutrition disorders) | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 21
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 36
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15
Dizziness (Nervous system disorders) | 16
Headache (Nervous system disorders) | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 32
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 13
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 16
Rash (Skin and subcutaneous tissue disorders) | 24
Vertigo (Ear and labyrinth disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 10
Chest pain (General disorders) | 10
Influenza like illness (General disorders) | 8
Bronchitis (Infections and infestations) | 8
Influenza (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 7
Viral upper respiratory tract infection (Infections and infestations) | 15
Blood creatinine increased (Investigations) | 7
Weight increased (Investigations) | 18
Hypokalaemia (Metabolism and nutrition disorders) | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8
Dysgeusia (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 14
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7

LIMITATIONS AND CAVEATS:
Part 1 analysis was not conducted as during the conduct of the study the RP2D was confirmed in study NP28761 (NCT01871805).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.